CLINICAL TRIAL: NCT04689048
Title: Characterization of Large Brain Metastases With 18F-Fluciclovine PET/CT Treated With Staged Stereotactic Radiosurgery
Brief Title: Assess Use of 18F-Fluciclovine for Patients With Large Brain Metastases Treated With Staged Stereotactic Radiosurgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-KOT-001
Record Dates: First submitted 2020-12-11; First posted 2020-12-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases, Adult; Brain Metastases; Brain Cancer
Keywords: brain; brain metastases; brain metastases, adult; brain cancer; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-site, single-arm, phase 1 proof-of-concept study to assess the potential clinical utility of 18F-fluciclovine PET/CT as a functional integral biomarker for patients with large brain metastases (>2 cm) treated with Staged Stereotactic Radiosurgery (SSRS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/CT, MRI (Other): In total, three 18F-fluciclovine PET/CT brain scans (pre-, interim-, and post-treatment) will be performed according to the study calendar. Generic name is Axumin and will be administered as an intravenous bolus. May administer diluted or undiluted. The maximum volume of undiluted 18F-fluciclovine is 5 mL. After administration, flush with normal saline to ensure full delivery of the dose.
  Interventions: Drug: 18F fluciclovine

INTERVENTIONS:
Drug: 18F fluciclovine — Patients will receive a standard 5 millicuries dose of 18F-fluciclovine intravenously as a bolus injection. They will be required to fast for at least four hours prior to 18F-fluciclovine injection. Patients will be positioned for PET/CT brain imaging and will be injected with 18F-fluciclovine immediately prior to PET data acquisition. PET data will be collected in list mode up to 25 minutes post-injection. PET images will be reconstructed in two ways: as a standard static image of data acquired between 10 to 20 minutes post-injection, and as a dynamic series of four 5-minute frames between 5 to 25 minutes post-injection to allow for motion assessment and correction and time-dependent observations.
  Other Names: Axumin

SUMMARY:
The spread of cancer to the brain is referred to as brain metastases. Brain metastases are a common complication of cancer. This study is being done to determine whether the use of a new imaging agent, 18F-fluciclovine, is able to detect which patients are responding to radiation therapy. In addition, this study will look at the changes of the treated brain metastases using this imaging agent over time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years
2. Performance status, Eastern Cooperative Oncology Group 0-2
3. Confirmed diagnosis of brain metastases with at least one untreated lesion >2 cm in maximum diameter
4. Plan for SSRS per the treating team
5. For women of childbearing potential, a negative serum pregnancy test within 14 days of registration is required
6. For females of reproductive potential: use of highly effective contraception for at least 4 weeks prior to screening and agreement to use such a method during study participation and for an additional 1 week after post-treatment 18F-fluciclovine positron emission tomography/computerized tomography

Exclusion Criteria:

1. Prior anaphylactic reaction to 18F-fluciclovine
2. Evidence of leptomeningeal disease
3. Prior whole-brain radiation therapy
4. Contraindication to MRI (e.g., due to safety reasons, such as presence of a pacemaker)
5. Females pregnant at the expected time of 18F-fluciclovine administration
6. Females who are expecting to be breastfeeding at the time of 18F-fluciclovine and unwilling to stop breast-feeding for 24 hours. Temporary cessation of breastfeeding 24 hours after the time of imaging is allowed
7. Major medical illness or psychiatric/cognitive impairments, which in the investigator's opinion, will prevent completion of protocol therapy and/or preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in sensitivity for PET/CT | through study completion, an average of 1 year
  Calculate the sensitivity of pre-treatment 18F-fluciclovine PET/CT to identify brain metastases >2 cm treated with SSRS.
Change in sensitivity for MRI | through study completion, an average of 1 year
  To calculate the sensitivity of pre-treatment contrast-enhanced MRI.
Change in the standardized uptake value (SUV) parameters | through study completion, an average of 1 year
  To identify a change in the standardized uptake value (SUV) parameters (SUVpeak, SUVmean, and SUVmax) for the 18F-fluciclovine PET/CT scans.

SECONDARY OUTCOMES:
Compare change of SUV metrics of 18F-fluciclovine PET | baseline
  To calculate the pre-, interim-, and post-treatment SUV metrics of 18F-fluciclovine PET uptake
Compare change of SUV metrics of contrast-enhanced MRI | baseline
  To calculate the percent change in lesion volume on contrast-enhanced MRI (∆MRIvolume).

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh R Kotecha, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125
- See also: Miami Cancer Institute website — http://baptisthealth.net/cancer-care/home